CLINICAL TRIAL: NCT02618629
Title: A Phase I Mass Balance and Metabolism Study of 14C-Z-215 in Healthy Male Volunteers
Brief Title: Mass Balance and Metabolism Study of 14C-Z-215
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Z215-03
Record Dates: First submitted 2015-11-27; First posted 2015-12-01 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14C-Z-215 (Experimental)
  Interventions: Drug: 14C-Z-215

INTERVENTIONS:
Drug: 14C-Z-215 — Single oral dose of 20mg Z-215 and 14C-Z-215 solution

SUMMARY:
The aim of this Phase I study is to determine the absorption, metabolism, and excretion of 14C-Z-215 in healthy male subjects following a single oral administration at a therapeutically relevant dose level (20 mg).

ELIGIBILITY:
Inclusion Criteria:

* Any race/ethnic origin
* Subjects will have a body mass index (BMI) between 18.5 and 30.0 kg/m2
* Subjects will have a body weight between 50 and 110 kg
* Subjects will have given their written informed consent to participate in the study, and to abide by the study restrictions.

Exclusion Criteria:

* Subjects who have a significant history of drug allergy, as determined by the Investigator.
* Subjects who have serum hepatitis or are carriers of the hepatitis B surface antigen (HBsAg) or the hepatitis C antibody.
* Subjects who have a positive result for the test for human immunodeficiency virus (HIV) antibodies.
* Subjects who are exposed to radiation as a result of their occupation.
* Subjects who, in the opinion of the Investigator, should not participate in this study.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Mass balance recovery of total radioactivity concentration in plasma, red blood cells and whole blood | Predose,15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours postdose
Concentration of Z-215 in plasma | Predose,15 and 30 minutes, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 14, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours postdose
Mass balance recovery of total radioactivity in urine | Predose, 0 to 6, 6 to 12, 12 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, 144 to 168, 168 to 192, 192 to 216, 216 to 240 hours postdose, Day 15 (336 hours postdose), Day 19 (432 hours postdose), Day 23 (528 hours postdose)
Mass balance recovery of total radioactivity in faecal | Predose, 0 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120, 120 to 144, 144 to 168, 168 to 192, 192 to 216, 216 to 240 hours postdose, Day 15 (336 hours postdose), Day 19 (432 hours postdose), Day 23 (528 hours postdose)

CONTACTS AND LOCATIONS:
Locations (1):
- UK, United Kingdom